CLINICAL TRIAL: NCT02259504
Title: COAST: Coiling of Aneurysms Smaller Than 5mm With Hypersoft® and Hydrogel Coils
Acronym: COAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PRO00035000
Record Dates: First submitted 2014-07-31; First posted 2014-10-08 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Small Intracranial Aneurysms
Keywords: aneurysms
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: PHASE 1- HyperSoft® 3D and HyperSoft® Helical Coils — Framing with HyperSoft® 3D or any FDA-approved bare platinum coil. Must fill and finish the the aneurysm with HyperSoft® 3D and/or HyperSoft® helical coils.
Other: PHASE 2 - HydroSoft® 3D and HydroSoft® Helical Coils — Framing with HydroFrame® or HydroSoft® 3D coils. Must fill the aneurysm with HydroFrame®, HydroSoft® (3D and/or Helical), and/or HydroFill® Coils and finish with HydroSoft® (3D and/or Helical) Coils.

SUMMARY:
This is a prospective, single-arm, multi-center post-marketing Study. The Study will commence as a single phase, with an optional second phase to follow at the discretion of the sponsor. Up to 300 eligible Subjects with small (< 4.9 mm) intracranial aneurysms, who consent to Study participation, will be treated in Phase 1 with MicroVention HyperSoft® 3D and HyperSoft® Helical coils with or without balloon remodeling or stent assistance at the discretion of the treating physician. The operator, at his/her discretion, may choose to frame the aneurysm with HyperSoft® 3D or any other bare metal coil but must finish the remainder of the aneurysm with HyperSoft® 3D and/or HyperSoft® Helical coils. At the discretion of the sponsor, additional patients, up to 300 patients total for the overall Study, with eligible aneurysms will be enrolled into Phase 2. In Phase 2, the aneurysm must be framed with a HydroFrame® or HydroSoft® 3D coil and filled/finished primarily with hydrogel coils. The intent to treat is to frame, fill and finish with all hydrogel coils. However, at the discretion of the treating physician, a bare platinum coil may be used to fill or finish, as long as a minimum of 50% (in total coil length) of hydrogel coils are used. Data will be collected on immediate and post-treatment angiographic occlusion rates (RRGS), new peri-procedural imaging-confirmed hemorrhage or ischemic stroke, neurological morbidity and mortality rates, recurrence rates, bleeding rates, retreatment rates, serious adverse events, >150 day angiographic occlusion rates (RRGS) and occlusion status. This will serve to establish the acute and sustained efficacy of EVT of small intracranial aneurysms with the specified microcoils, aided by balloon and/or stent remodeling where appropriate.

DETAILED DESCRIPTION:
1.0 INTRODUCTION 1.1 Background Intracranial aneurysms (IAs) are common cerebrovascular abnormalities. The prevalence of IAs has been reported to be 0.8-2.0% of the population. [1-3] The most common presentation of IAs is subarachnoid hemorrhage (SAH), the annual incidence of which varies by geographic region from 10 to 20 per 100,000. [4 5] SAH is a devastating injury with a case-fatality rate of 51% [5]. Nearly half of its survivors are functionally incapacitated [6].

There is limited data on the natural history of small intracranial aneurysms. According to the International Study of Unruptured Intracranial Aneurysms, the risk of spontaneous aneurysm rupture is related to aneurysm size and location. ISUIA found aneurysms < 10 mm in diameter, as opposed to aneurysms 10-24 mm and >25 mm, had relative risks of rupture of 11.6 and 59, respectively. Further follow-up from this cohort showed 5-year bleeding risks of 0%, 2.6%, 14.5%, and 40% for aneurysms less than 7 mm, 7--12 mm, 13--24 mm, and 25 mm or greater, respectively. Many other authors (Juvela 2000 and Weir 2002) also suggest the risk of small aneurysm rupture is relatively low. The Sapporo SAH Study group suggests that while the overall rupture risk of small aneurysms is low, the aneurysm size ratio is a strong predictor of aneurysm rupture in small (<5mm) intracranial aneurysms [7]. However, some authors and unpublished data (MUSC) demonstrate that approximately one-third of all ruptured aneurysms are less than 4 mm in size.

Endovascular coiling of intracranial aneurysms has been shown to be safe and efficacious in the treatment of intracranial aneurysms. The International Subarachnoid Aneurysm Trial (ISAT) has shown that endovascular coiling can reduce morbidity and mortality compared to clipping of aneurysms in the setting of SAH. [8]. The goal of endovascular coiling is to prevent rupture or rebleeding by isolating an aneurysm from the normal blood circulation without narrowing the parent vessel.

A main concern of endovascular treatment is the long-term durability of treatment, that is to say that it is possible for the aneurysm to recanalize (recur) after it has been treated with coils [9]. Some factors in recanalization are incomplete initial occlusion, large aneurysm size, ruptured aneurysm, partially thrombosed aneurysm, and compaction of the coil mass within the aneurysm [9 10]. In a Study by Nguyen [11], incomplete initial aneurysm occlusion, rupture and large aneurysm size were all associated with significant recanalization. Johnston [12] concluded the degree of occlusion after initial treatment to be a strong predictor of the risk of subsequent rupture, which justified attempts to completely occlude aneurysms. Two series of small unruptured intracranial aneurysms [13 14] found recurrence rates between 5.9% and 16.9% with retreatment rates of 1.7% and 2.9%. The majority of retreatments were in small wide necked aneurysms. However, the recurrence rates of small aneurysms is much less than those of large aneurysms (71% vs 35%) [15].

The other main concern with the treatment of small aneurysms (less than 4 mm) is safety, namely the concern of intraprocedural rupture or thromboembolic events. The ATENA Study showed that the risk of intraprocedural aneurysm rupture was significantly higher in small aneurysms (3.7% for 1-6 mm vs 7% for 7-15 mm; p= 0.008). The rate of failure of EVT was significantly higher in very small unruptured aneurysms compared to larger aneurysms (13.7% vs 3.3% respectively). This is likely related to several factors. Microcatheterization of the aneurysm sac may be challenging due to aneurysm size and placing even the smallest coils, maybe challenging in small aneurysms. In the same series as above [13 14], a 10.4% overall procedural complication rate was found. There were 24 embolic events, 11 coil protrusions and 4 aneurysm ruptures, while Oishi found a 3.8% thromboembolic event rate and a 1.4% risk of aneurysm rupture. Nguyen et al reported an intraprocedural rupture rate of 11.7% in aneurysms less than 3 mm in diameter [16]. In a meta-analysis, Brinjikji et al found a procedural rupture rate of 8.3% in small aneurysms while Spiotta et al demonstrated a 13.5% rate of intraprocedural rupture in ruptured aneurysms less than 4 mm [17] Other studies have found morbidity and mortality rates that range from 0.8%-7% and 0-1.4% [13 14 18]. The introduction of the Microvention HyperSoft® 3D line of coils with sizes from 1 to 5mm may help reduce these historical risks of failure to treat and intraprocedural rupture. The complex shape of the coils may allow for stable framing of the aneurysms followed by dense packing of the aneurysm sac and neck, therefore preventing recurrence. The softness of the coils may allow for increased confidence and safety when treating these aneurysms, which may be expressed as a reduction of intraprocedural complications.

1.2 Pathophysiology and Prevalence of Aneurysms A cerebral or intracranial aneurysm is a focal dilation of an artery in the brain that results from a weakening of the inner muscular layer (the intima) of a blood vessel wall. The pathogenesis of intracranial aneurysms remains incompletely understood. Most aneurysms arise sporadically but occasionally they may be: dissecting (resulting from a luminal endothelial tear), traumatic (usually within 2-3 weeks after severe head injury) or mycotic (as a result of embolism of infected material). Aneurysm etiology is multifactorial, including congenital medial arterial wall defects, degenerative changes, and accruing hemodynamic stress, particularly at sites of turbulent blood flow. Contributing factors include connective tissue disorders, hypertension, anatomy variations, atherosclerosis, trauma, mycosis, and tumors. Epidemiological studies have already identified aneurysm-specific risk factors such as size and location, as well as patient-specific risk factors, such as age (higher in adults), sex (higher in females), and presence of medical comorbidities, such as hypertension. In addition, exposure to certain environmental factors such as smoking has been shown to be important in the formation of IA. Furthermore, substantial evidence proves that certain loci contribute genetically to IA pathogenesis. Genome-wide linkage studies using relative pairs or rare families that are affected with the Mendelian forms of IA have already shown genetic heterogeneity of IA, suggesting that multiple genes, alone or in combination, are important in the disease pathophysiology [19].

Aneurysm wall thickness varies throughout the sac. The thickness is greatest at the neck and least at the fundus. Compared to small aneurysms, calcification and atheromas are more commonly seen in large aneurysms. Macrophages, present in all stages of atherosclerosis, secrete lytic enzymes (e.g., elastases, collagenases, metalloproteases), lead to the destruction of connective tissue and erosion of the arterial wall. Smooth muscle cell apoptosis and elastin/collagen fiber reconstruction mechanisms contribute to vessel wall weakening [20]. The weakening of aneurysm walls has been demonstrated in histological studies that found degeneration of endothelial cells and internal elastic lamina and thinning of the medial layer [21]. Aneurysm wall tensions and stressors have been noted to be an important contributor to growth, remodeling and rupture in aneurysms. Focal turbulence and discontinuity of the normal architecture at vessel bifurcations may account for the propensity of saccular aneurysm formation [22].

The frequency of cerebral aneurysms is difficult to ascertain because of variation in the definitions of the size of aneurysm and modes of detection. Autopsy series cite prevalences of 0.2-7.9%. Prevalence ranges from 5-10%, with unruptured aneurysms accounting for 50% of all aneurysms. Pediatric aneurysms account for only 2% of all cerebral aneurysms. In the United States, the incidence of ruptured aneurysms is approximately 12 per 100,000 individuals or 30,000 annual cases of aneurysmal SAH. The frequency of cerebral aneurysms has not declined in recent years. [22] Saccular (berry) aneurysms constitute 90% of all cerebral aneurysms and are usually located at the major branch points of large arteries. Saccular aneurysms frequently rupture into the subarachnoid space, accounting for 70-80% of spontaneous subarachnoid hemorrhage. Annually, 15,000 American patients have SAH from aneurysms with a maximum diameter <7 mm and consequently experience irreparable morbidity and severe mortality. The majority of their aneurysms were unruptured, single, asymptomatic, and even smaller at some point before rupture [23]. Fusiform or arteriosclerotic aneurysms are elongated outpouchings of proximal arteries that account for 7% of all cerebral aneurysms and infectious or mycotic aneurysms usually situated peripherally comprise 0.5% of all cerebral aneurysms. Small aneurysms are less than 10 mm in diameter. Larger aneurysms are 10-25 mm and giant aneurysms are greater than 25 mm in diameter [24]. About 80-90% of the aneurysms are small and only 10-20% are large and giant [5].

Both ruptured and unruptured aneurysms are candidates for endovascular therapy. The natural history of unruptured intracranial aneurysms is still unclear and is influenced by many factors such as previous subarachnoid hemorrhage from another aneurysm, history of cigarette smoking, coexisting medical conditions, and aneurysm characteristics such as size, location, and morphology [25]. In a Study of the natural history of aneurysms to determine the risk of rupture, Juvela [26] followed 142 patients with 181 unruptured aneurysms for a mean of 13.9 years (range 0.8 - 30 years) to death or subarachnoid hemorrhage. The annual rupture rate was 1.4%. The median diameter of the aneurysm followed was 4 mm at diagnosis. Fourteen of the intracranial hemorrhages (ICH) were fatal; the authors concluded that unruptured aneurysms should be treated if technically feasible irrespective of size.

1.3 Treatment options for intracranial aneurysms The wide availability and use of noninvasive imaging has increased the frequency of incidental discovery of intracranial aneurysms. There are two broad categories of intracranial aneurysms: those that have ruptured, creating subarachnoid hemorrhage and those that are unruptured. Subarachnoid hemorrhage from aneurysm rupture is a devastating event. It is estimated that about 40% of individuals whose aneurysm has ruptured do not survive the first 24 hours: up to another 25% die from complications within 6 months. Early diagnosis and treatment are important. [27] Aneurysm treatments include medical, surgical and endovascular therapies. Medical therapy involves general supportive measures and prevention of complications for individuals who are in the periprocedural period or are poor surgical candidates and includes: control of hypertension, calcium channel blockers, prevention of seizures and antibiotic therapy for those presenting with infectious aneurysms. In the microsurgical approach, a section of the skull is removed. The brain tissue is then spread apart to reveal the aneurysm and a small metal clip is placed at the base of the aneurysm to block the flow of blood. Alternative microsurgical techniques involve proximal or Hunterian ligation, wrapping of the aneurysm or trapping (i.e., a combination of proximal and distal vessel occlusion). [22] Endovascular therapy (EVT) involves insertion of a catheter into the femoral artery in the patient's leg and navigating it though the vascular system into the head and aneurysm. Once there, several treatment options are available: detachable coils may be deployed within the aneurysm to occlude it from the parent artery blood flow, this may be done alone or by using an adjunctive technique such as balloon remodeling or intracranial stenting of the parent artery. In balloon remodeling, a temporary occlusion balloon is inflated across the neck of the aneurysm while the coils are introduced. The balloon functions to prevent the prolapse of coils into the parent vessel. Although the temporary occlusion balloons provide support for the coils during their introduction, sometimes the coil can prolapse into the parent artery immediately after balloon deflation [28]. Also very wide-necked or irregular shaped aneurysms may lack a neck structure making coil placement difficult or impossible. These aneurysms may have an intracranial stent placed in the parent artery crossing the neck of the aneurysm. The coils are then introduced through the stent in order to help jail them within the aneurysm. Parent vessel occlusion, although not as common as aneurysm coiling is performed mostly on fusiform and acute dissecting arteries and involves the complete occlusion of the parent vessel with coils and sometimes embolic liquid.

Embolization with detachable coils is a safe and effective treatment of brain aneurysms. The 1-year results of the ISAT Study [29] of endovascular coiling of aneurysms (considered suitable for both neurosurgical clipping and endovascular coiling) yielded a significant advantage over neurosurgical clipping in terms of death and severe disability. Of patients allocated to endovascular treatment, 250 of 1063 (23.5%) were dead or dependent at 1 year compared with 326 of 1055 (30.9%) patients allocated to neurosurgical clipping. As such, the absolute risk reduction was calculated as 7.4% (95% CI: 3.6-11.2; P = .0001) in favor of endovascular treatment. Because of this significant difference between coiling and clipping, treatment of patients with a ruptured intracranial aneurysm changed significantly over the past years, particularly in Europe. In many centers, coiling has become the method of choice when both coiling and clipping are considered suitable in the individual patient.

At 5 years, 11% (112 of 1046) of the patients in the endovascular group and 14% (144 of 1041) of the patients in the neurosurgical group had died. The risk of death at 5 years was significantly lower in the coiling group than in the clipping group [8].

Although endovascular coiling has been shown to be a safe and effective treatment, some of these same patients require repeat treatment for recurrence of an aneurysm [30 31]. Published series regarding mid and long-term clinical outcome and follow up angiographic findings confirm that recanalization may occur in up to 33% of treated patients, which also tends to increase in the aneurysms with wider necks and larger sizes [2 30 32 33]. In the case of coiled aneurysms, large aneurysms are more likely to recur than smaller ones and ruptured aneurysms are more likely to recur than unruptured ones [11 30].

Over the last decade, there have been significant improvements of the endovascular techniques and the development of a wide range of devices including 3-D coils, spherical coils, and complex coils. The introduction of balloon and stent remodeling techniques resulted in further expansion of the devices and techniques available to neurointerventionalists, and made EVT possible for greater percentage of patients. Enhancement of platinum coil thrombogenicity has been attempted by surface modifications using Dacron® fibers, bioabsorbable polymers (Cerecyte® coil, Codman/Micrus Endovascular; Matrix®coil, Boston Scientific) or hydrogel coatings (HydroCoil®, MicroVention). The use of non adhesive embolic agents such as Onyx® (ev3) for aneurysm embolization has proven to be an occlusive method that, in some patients, completely fills and conforms to the unique geometry of the aneurysm cavity, resulting in complete aneurysm obliteration. A relatively new technique being used is Parent Vessel Reconstruction using stents (Neuroform® microstent Boston Scientific, Enterprise™ Codman®, Pipeline Embolization Device, Covidien) not just to coil the aneurysm but to change the parent vessel configuration, redirect the flow of blood to help reduce the wall shear stress on the aneurysm and to promote tissue growth over the neck of the aneurysm.

2.0 STUDY OBJECTIVES The primary objective of this post-marketing Study is to assess the clinical and imaging outcomes in the endovascular treatment of small (≤ 4.9 mm) intracranial aneurysms utilizing the HyperSoft® 3D and HyperSoft® Helical coils (or HydroFrame®, HydroFill® and HydroSoft® (3D and Helical) coils in Phase 2) specifically designed for the treatment of small aneurysms. The neck of the aneurysm may be protected during coiling with a balloon or stent indicated for use in the neurovasculature.

It is hypothesized that framing, filling and neck finishing using HyperSoft® 3D, HydroFrame®, HydroSoft® 3D and HyperSoft® Helical coils, aided by balloon remodeling or stent assistance where appropriate, will yield better occlusion rates, may lower recanalization and retreatment rates and be safer (reduce intraprocedural aneurysm rupture rates) compared to historical data using earlier generation technology.

2.1 Primary Endpoints

* Efficacy: Raymond-Roy grading scale (RRGS) of 2 or better occlusion on follow up angiography performed >150 days post embolization, not requiring retreatment
* Safety: Freedom from imaging-confirmed new post-procedural hemorrhage and ischemic stroke associated with a 4-point worsening in NIHSS within 48 hours of aneurysm treatment or any new aneurysmal SAH secondary to treated aneurysm 2.2 Secondary Endpoints
* Any neurological morbidity and mortality (evaluated at time of >150-day angiographic follow up)
* Bleeding rate of target aneurysms, including rebleeding of target ruptured aneurysms (at one year)
* Recurrence rate/recanalization (evaluated at time of >150-day angiographic follow up)
* Retreatment rate (at one year)

ELIGIBILITY:
Inclusion Criteria

Candidates for this Study must meet all of the following criteria to be enrolled in the Study:

1. Subject age ≥ 18 and ≤ 80 with a diagnosis of ruptured or unruptured saccular intracranial aneurysm judged suitable for selective endovascular treatment by coil occlusion
2. Aneurysm size [largest measurement from the cross sectional images to determine overall aneurysm size, not just the lumen, and including any thrombosed portions] ≤ 4.9 mm
3. If ruptured aneurysm: Hunt and Hess 0-3
4. If unruptured aneurysm: Subject grade Modified Rankin Scale mRS 0 - 2 The investigator believes the aneurysm is appropriate for the designated Phase coiling paradigm. (Phase 1: Frame, fill and finish with MicroVention HyperSoft® 3D and/or HyperSoft® Helical coils). The operator at his discretion may frame with any bare metal framing coil but the remainder of the coils must be HyperSoft® 3D or HyperSoft® Helical coils. Phase 2: Frame with MicroVention HydroFrame® or HydroSoft® 3D coils and fill/finish with sufficient hydrogel coils to ensure 50% hydrogel by length. The intent to treat is to frame, fill and finish with all hydrogel coils. However, at the discretion of the treating physician, a bare platinum coil may be used to fill or finish, as long as a minimum of 50% (in total coil length) of hydrogel coils are used.
5. Signed informed consent.

Exclusion Criteria

Candidates will be ineligible for enrollment in the Study if any of the following conditions apply:

1. Patient has more than one aneurysm requiring treatment in the current treatment session, and only one of those to be treated aneurysms fits the current Study inclusion criteria (i.e. if either (1) a patient has multiple aneurysms, but only one will be treated at enrollment; or (2) if two or more aneurysms are treated during the current treatment session and BOTH are able to be enrolled, then they remain eligible for the Study). Non-treated additional aneurysms may be treated after 30 days from the incident procedure with any coil type that the operator chooses, and, if eligible, those aneurysms may also be enrolled as an additional enrollment.
2. Prior treatment (surgical or endovascular) of the target aneurysm
3. Subject with social, medical, or psychological conditions that interfere with treatment and follow-up evaluation
4. Women who are pregnant or plan to become pregnant during the Study
5. Use of other modified coils (Matrix, HydroCoil® or fibered coils) - except Phase 2 as noted above in the inclusion criteria
6. Use (current or prior) of liquid embolic material in the treatment of the target aneurysm
7. Life expectancy less than 12 months
8. Presence of arteriovenous malformation or fistula
9. Presence of fusiform, mycotic, traumatic, dissecting or tumoral aneurysms in any location 10. Intended or planned aneurysm treatment by parent vessel occlusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2014-07; Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Imaging outcomes (occlusion results) of small intracranial aneurysms as defined by the raymond Roy Grading scale. | 48 hours
  To measure imaging outcomes of small (≤ 4.9 mm) intracranial aneurysms utilizing the HyperSoft® 3D (and HydroSoft® 3D, when commercially available) and HyperSoft® helical coils specifically designed for the treatment of small aneurysms.

SECONDARY OUTCOMES:
Neurological morbidity/mortality (degree of functionality) defined by the Modified Rankin Scale (mRS) | one year
  Measure any neurological morbidity/mortality (evaluated at time of >150-day angiographic follow up)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lena, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States